CLINICAL TRIAL: NCT01543035
Title: Phase III Prospective Multicentric Trial Evaluating Etravirine for HIV Infected Patients in Need of Lipid Lowering Drugs: the ETRALL Trial
Brief Title: Prospective Evaluation of Etravirine for HIV-infected Patients in Need of Lipid-lowering Drugs
Acronym: ETRALL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Calmy Alexandra (Other)
Collaborators: Janssen-Cilag A.G., Switzerland (Industry)
Responsible Party: Sponsor-Investigator, Calmy Alexandra, MD, PhD, HIV department Director, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETRALL DR3215
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infection
Keywords: HIV infection; lipid lowering drugs; etravirine; patient; statin treatment; EFV or boosted PI antiretroviral treatment
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etravirine switch (Experimental): Patients in need of lipid-lowering drug switched from boosted PI or EFV to Etravirine
  Interventions: Drug: stop statin and switch to an antiretroviral drug with less impact on lipid metabolism

INTERVENTIONS:
Drug: stop statin and switch to an antiretroviral drug with less impact on lipid metabolism — Switch from a boosted PI or efavirenz based ART regimen to etravirine 400 mg/day once daily for patients in need of lipid lowering drugs (statin) after one month wash out of statin

SUMMARY:
Dyslipidaemia, characterized by raised triglyceride and low-density lipoprotein (LDL) cholesterol and reduced high-density lipoprotein (HDL) cholesterol levels, is common in HIV-infected individuals, and has been associated with HIV infection itself and antiretroviral therapy (ART). These abnormalities are well-established markers of cardiovascular (CVD) risk in the general population. Studies have suggested an increased risk of CVD associated with ART exposure over and above that conveyed by traditional cardiovascular risk factors. In HIV population to reduce lipid parameters, the most usual clinical strategy remains to add a statin treatment.

Recent studies suggested ART switch can represent an interesting alternative to statins to reduce lipid plasma levels.

The purpose of this study is to evaluate the frequency with which the replacement of LPV/r (lopinavir/ritonavir), ATZ/r (atazanavir/ritonavir), DRV/r (darunavir/ritonavir) or EFV (efavirenz) by ETR (Etravirin) in dyslipidemic patients with suppressed viremia would obviate the necessity to administer statins.

A prospective, phase III study in which the statin treatment of dyslipidemic HIV patients on antiretroviral drugs (ARVs) will be interrupted during 4 weeks is proposed.

At week 4, patients qualifying for a lipid lowering drug (calculated LDL-C≥ 3mmol/L) will replace EFV, LPV/r, DRV/r or ATZ/r by ETR. The proportion of patients not qualifying anymore for a statin treatment at 12 weeks (i.e. after 8 weeks of ETR treatment) will be determined. Additionally, the lipid level changes will be assessed at 12 weeks. Inflammatory markers will be measured at baseline, at drug switch and at the end of the study

Study drug will be provided by the drug manufacturer (Janssen-Cilag, AG). Compliance for study drug will be done at week-4 and week-12, Returned study medication will be counted and the amount notified on the Case Report Form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* On statin treatment for at least 3 months (fluvastatin, simvastatin, pravastatin, rosuvastatin, or atorvastatin) for primary prevention of cardiovascular disease
* HIV Ribonucleic Acid (RNA) below 50 copies/mL, minimum duration 3 months
* On a stable (> 3 months) ARV treatment including at least one of the following drugs: LPV/r, ATZ/r, DRV/r, or EFV
* No previous virological escape or virological escape documented with a genotype at the time of failure only showing a K103M mutation.

Exclusion Criteria:

* Probability of cardiovascular complications of > 20% according to the Swiss GSLA ("Groupe de travail Lipide et Athérosclérose"/Swiss Atherosclerosis Association) guidelines
* Previous cardiovascular disease (including stroke)
* Known diabetes
* Known intolerance of ETR
* Presence of a documented drug mutation (excluding the K103M)
* Regimen including non-boosted ATZ
* Known hyperlipidemia before ARV initiation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients not qualifying anymore for statin treatment | 12 weeks

SECONDARY OUTCOMES:
fasting lipids changes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Calmy Alexandra, Md, PhD, Principal Investigator — University Hospital, Geneva
Locations (7):
- Switzerland (7):
  - Universitätsspital Basel Klinik für Infektiologie & Spitalhygiene, Basel
  - Inselspital PKT2B / Poliklinik für Infektiologie, Bern
  - HUG /Division des Maladies infectieuses Unité VIH/SIDA, Geneva
  - Hôpital Neuchâtelois - La Chaux-de-Fonds Service des Maladies infectieuses, La Chaux-de-Fonds
  - CHUV / Service des maladies infectieuses Médecine 2, Lausanne
  - Kantonsspital / Infektiologie und Spitalhygiene Departement Innere Medizin, Sankt Gallen
  - Universitätsspital Zürich Division of Infectious Diseases and Hospital Epidemiology Department of Internal Medicine, Zurich

REFERENCES:
- [Background] Riddler SA, Li X, Chu H, Kingsley LA, Dobs A, Evans R, Palella F, Visscher B, Chmiel JS, Sharrett A. Longitudinal changes in serum lipids among HIV-infected men on highly active antiretroviral therapy. HIV Med. 2007 Jul;8(5):280-7. doi: 10.1111/j.1468-1293.2007.00470.x. PMID 17561873
- [Background] Grunfeld C, Pang M, Doerrler W, Shigenaga JK, Jensen P, Feingold KR. Lipids, lipoproteins, triglyceride clearance, and cytokines in human immunodeficiency virus infection and the acquired immunodeficiency syndrome. J Clin Endocrinol Metab. 1992 May;74(5):1045-52. doi: 10.1210/jcem.74.5.1373735.
- [Background] Riddler SA, Smit E, Cole SR, Li R, Chmiel JS, Dobs A, Palella F, Visscher B, Evans R, Kingsley LA. Impact of HIV infection and HAART on serum lipids in men. JAMA. 2003 Jun 11;289(22):2978-82. doi: 10.1001/jama.289.22.2978. PMID 12799406
- [Background] Carr A, Samaras K, Burton S, Law M, Freund J, Chisholm DJ, Cooper DA. A syndrome of peripheral lipodystrophy, hyperlipidaemia and insulin resistance in patients receiving HIV protease inhibitors. AIDS. 1998 May 7;12(7):F51-8. doi: 10.1097/00002030-199807000-00003. PMID 9619798
- [Background] Mulligan K, Grunfeld C, Tai VW, Algren H, Pang M, Chernoff DN, Lo JC, Schambelan M. Hyperlipidemia and insulin resistance are induced by protease inhibitors independent of changes in body composition in patients with HIV infection. J Acquir Immune Defic Syndr. 2000 Jan 1;23(1):35-43. doi: 10.1097/00126334-200001010-00005. PMID 10708054
- [Background] Thiebaut R, Daucourt V, Mercie P, Ekouevi DK, Malvy D, Morlat P, Dupon M, Neau D, Farbos S, Marimoutou C, Dabis F. Lipodystrophy, metabolic disorders, and human immunodeficiency virus infection: Aquitaine Cohort, France, 1999. Groupe d'Epidemiologie Clinique du Syndrome d'Immunodeficience Acquise en Aquitaine. Clin Infect Dis. 2000 Dec;31(6):1482-7. doi: 10.1086/317477. Epub 2000 Nov 29. PMID 11096016
- [Background] Wand H, Calmy A, Carey DL, Samaras K, Carr A, Law MG, Cooper DA, Emery S; INITIO Trial International Coordinating Committee. Metabolic syndrome, cardiovascular disease and type 2 diabetes mellitus after initiation of antiretroviral therapy in HIV infection. AIDS. 2007 Nov 30;21(18):2445-53. doi: 10.1097/QAD.0b013e3282efad32. PMID 18025881
- [Background] Friis-Moller N, Sabin CA, Weber R, d'Arminio Monforte A, El-Sadr WM, Reiss P, Thiebaut R, Morfeldt L, De Wit S, Pradier C, Calvo G, Law MG, Kirk O, Phillips AN, Lundgren JD; Data Collection on Adverse Events of Anti-HIV Drugs (DAD) Study Group. Combination antiretroviral therapy and the risk of myocardial infarction. N Engl J Med. 2003 Nov 20;349(21):1993-2003. doi: 10.1056/NEJMoa030218. PMID 14627784
- [Background] DAD Study Group; Friis-Moller N, Reiss P, Sabin CA, Weber R, Monforte Ad, El-Sadr W, Thiebaut R, De Wit S, Kirk O, Fontas E, Law MG, Phillips A, Lundgren JD. Class of antiretroviral drugs and the risk of myocardial infarction. N Engl J Med. 2007 Apr 26;356(17):1723-35. doi: 10.1056/NEJMoa062744. PMID 17460226
- [Background] Carey D, Amin J, Boyd M, Petoumenos K, Emery S. Lipid profiles in HIV-infected adults receiving atazanavir and atazanavir/ritonavir: systematic review and meta-analysis of randomized controlled trials. J Antimicrob Chemother. 2010 Sep;65(9):1878-88. doi: 10.1093/jac/dkq231. Epub 2010 Jun 16. PMID 20554568
- [Background] Sension M, Andrade Neto JL, Grinsztejn B, Molina JM, Zavala I, Gonzalez-Garcia J, Donnelly A, Phiri P, Ledesma E, McGrath D; 067 Study Group. Improvement in lipid profiles in antiretroviral-experienced HIV-positive patients with hyperlipidemia after a switch to unboosted atazanavir. J Acquir Immune Defic Syndr. 2009 Jun 1;51(2):153-62. doi: 10.1097/QAI.0b013e3181a5701c. PMID 19346966
- [Background] Nguyen A, Calmy A, Delhumeau C, Mercier IK, Cavassini M, Fayet-Mello A, Elzi L, Genne D, Rauch A, Bernasconi E, Hirschel B; Swiss HIV Cohort Study. A randomized crossover study to compare efavirenz and etravirine treatment. AIDS. 2011 Jan 2;25(1):57-63. doi: 10.1097/QAD.0b013e32833f9f63. PMID 21076278
- [Background] Ruxrungtham K, Pedro RJ, Latiff GH, Conradie F, Domingo P, Lupo S, Pumpradit W, Vingerhoets JH, Peeters M, Peeters I, Kakuda TN, De Smedt G, Woodfall B; TMC125-C227 study group. Impact of reverse transcriptase resistance on the efficacy of TMC125 (etravirine) with two nucleoside reverse transcriptase inhibitors in protease inhibitor-naive, nonnucleoside reverse transcriptase inhibitor-experienced patients: study TMC125-C227. HIV Med. 2008 Nov;9(10):883-96. doi: 10.1111/j.1468-1293.2008.00644.x. Epub 2008 Sep 14. PMID 18795960
- [Background] Spencer FA, Allegrone J, Goldberg RJ, Gore JM, Fox KA, Granger CB, Mehta RH, Brieger D; GRACE Investigators. Association of statin therapy with outcomes of acute coronary syndromes: the GRACE study. Ann Intern Med. 2004 Jun 1;140(11):857-66. doi: 10.7326/0003-4819-140-11-200406010-00006. PMID 15172899
- [Background] McGowan MP; Treating to New Target (TNT) Study Group. There is no evidence for an increase in acute coronary syndromes after short-term abrupt discontinuation of statins in stable cardiac patients. Circulation. 2004 Oct 19;110(16):2333-5. doi: 10.1161/01.CIR.0000145118.55201.15. Epub 2004 Oct 11. PMID 15477411
- [Derived] Ciaffi L, Cavassini M, Genne D, Delhumeau C, Spycher Elbes R, Hill A, Wandeler G, Fehr J, Stoeckle M, Schmid P, Hirschel B, Montecucco F, Calmy A; Swiss HIV Cohort Study. Switch to etravirine for HIV-positive patients receiving statin treatment: a prospective study. Eur J Clin Invest. 2015 Jul;45(7):720-30. doi: 10.1111/eci.12464. PMID 25989829